CLINICAL TRIAL: NCT07134127
Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effect of IBI3032 in Participants
Brief Title: A Study of IBI3032 in Chinese Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Innovent Biologics Technology Limited (Shanghai R&D Center) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CIBI3032T001
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Single dose1 of IBI3032 administered orally. (Experimental): dose1 IBI3032
  Interventions: Drug: IBI3032
- Single dose4 of placebo administered orally. (Placebo Comparator): dose4 placebo
  Interventions: Drug: placebo
- Single dose4 of IBI3032 administered orally. (Experimental): dose4 IBI3032
  Interventions: Drug: IBI3032
- D1:Single dose3-1 of placebo administered orally. D9:Single dose3-1 of placebo administered orally. (Active Comparator): D1: Fasted administer D9:Administer after meal
  Interventions: Drug: placebo
- Single dose2 of IBI3032 administered orally. (Experimental): dose2 IBI3032
  Interventions: Drug: IBI3032
- D1:Single dose3-2 of placebo administered orally. D9:Single dose3-2 of placebo administered orally. (Active Comparator): D1:Administer after meal D9: Fasted administer
  Interventions: Drug: placebo
- D1:Single dose3-2 of IBI3032 administered orally. D9:Single dose3-2 of IBI3032 administered orally. (Experimental): D1:Administer after meal D9: Fasted administer
  Interventions: Drug: IBI3032
- D1:Single dose3-1 of IBI3032 administered orally. D9:Single dose3-1 of IBI3032 administered orally. (Experimental): D1: Fasted administer D9:Administer after meal
  Interventions: Drug: IBI3032
- Single dose1 of placebo administered orally. (Placebo Comparator): dose1 placebo
  Interventions: Drug: placebo
- Single dose2 of placebo administered orally. (Placebo Comparator): dose2 placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Placebo (without active ingredients) (cohort1, 2,4) Method of administration: oral, fasted administration. Placebo (without active ingredients) (cohort3) Method of administration: oral, administration after meal.
  Arms: D1:Single dose3-1 of placebo administered orally. D9:Single dose3-1 of placebo administered orally.; D1:Single dose3-2 of placebo administered orally. D9:Single dose3-2 of placebo administered orally.; Single dose1 of placebo administered orally.; Single dose2 of placebo administered orally.; Single dose4 of placebo administered orally.
Drug: IBI3032 — IBI3032: (cohort1, 2,4) Method of administration: oral, fasted administration. IBI3032: (cohort3) Method of administration: oral, administration after meal.
  Arms: D1:Single dose3-1 of IBI3032 administered orally. D9:Single dose3-1 of IBI3032 administered orally.; D1:Single dose3-2 of IBI3032 administered orally. D9:Single dose3-2 of IBI3032 administered orally.; Single dose1 of IBI3032 administered orally.; Single dose2 of IBI3032 administered orally.; Single dose4 of IBI3032 administered orally.

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase I clinical study evaluating the safety, tolerability, PK and food effect of a single dose of IBI3032 in healthy participants. This is a single ascending dose (SAD) study. Approximately 40 healthy participants are expected to be enrolled in this study. The screening period is 4 weeks. Eligible participants will be divided into 4 cohorts. Cohort1,2,4 consisted of 8 healthy participants who will be randomized in a 6:2 ratio to receive a single dose of IBI3032 or placebo. The safety follow-up period is 15 days. Cohort 3 consisted of 16 participants used a two-cycle, double-crossover design, who were randomly divided into four groups at a ratio of 3:1:3:1: Cohort 3-1-IBI3032, cohort 3-1-placebo, cohort 3-2-IBI3032, and cohort 3-2-placebo, each subject underwent two cycles of the trial. In cohort 3-1, the first cycle was given on fasted administration, and the second cycle was given after breakfast. In cohort 3-2, the first cycle was administered after breakfast intake, and the second cycle was administered fasted. The washout period for cohort 3-1 and cohort 3-2 was 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females, as determined by medical history
* Have safety laboratory results within normal reference ranges

Exclusion Criteria:

* Have known allergies toIBI3032， glucagon-like peptide-1 (GLP-1) analogs, related compounds
* Abnormal electrocardiogram (ECG) at screening
* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-29 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One Serious Adverse Event(s) Considered by the Investigator to be Related to Study Drug | (Cohoet1,2,4) Baseline up to Day 15 (Cohoet3) Baseline up to Day 15
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug | (Cohoet1,2,4) Baseline up to Day 15 (Cohoet3) Baseline up to Day 15
  A summary of other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with adverse events (AEs) | (Cohoet1,2,4) Baseline up to Day 15 (Cohoet3) Baseline up to Day 15
  An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

SECONDARY OUTCOMES:
Under the Serum Concentration-time Curve (AUC) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
maximum concentration (Cmax) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
time to maximum concentration (Tmax) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
clearance (CL) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
apparent volume of distribution (V) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.
elimination half-life (T1/2) of IBI3032 | Predose up to 168 hours postdose
  To evaluate the pharmacokinetic (PK) characteristics of a single dose of IBI3032 in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- The Frist Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China